CLINICAL TRIAL: NCT02807298
Title: 4% Articaine and 2% Lidocaine by Intraligamentary Technique in Irreversible Pulpitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. D. Y. Patil Dental College & Hospital (Other)
Responsible Party: Principal Investigator, Soumya Shetty, Dr., Dr. D. Y. Patil Dental College & Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DYPDCH/IEC-SS/18/2014
Record Dates: First submitted 2016-06-09; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Irreversible Pulpitis
Keywords: Intarligamentary; Articaine; Lidocaine
MeSH Terms: interventions — Lidocaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 2% Lignocaine (lidocaine) (Active Comparator): Intraligamentary injections of 1.8 ml of lidocaine and 1:100,000 epinephrine (adrenaline)
  Interventions: Drug: 2% Lignocaine; Drug: Epinephrine
- 4% Articaine (Experimental): intraligamentary injections of 0.9 ml of 4%articaine and 1:100,000 epinephrine (adrenaline)
  Interventions: Drug: 4%articaine; Drug: Epinephrine

INTERVENTIONS:
Drug: 4%articaine — intraligamentary injections of 0.9 ml of 4%articaine and 1:100,000 epinephrine
  Arms: 4% Articaine
Drug: 2% Lignocaine — Intraligamentary injections of 1.8 ml of lidocaine and 1:100,000 epinephrine
  Arms: 2% Lignocaine (lidocaine)
Drug: Epinephrine — Intraligamentary injections of 1.8 ml of lidocaine and 1:100,000 epinephrine

SUMMARY:
This study compared the anesthetic efficacy between Lignocaine and articaine administering it intraligamentarly using ligajet in twenty five female patients having irreversible pulpitis on bilateral mandibular molars. At 5minutes of post injection, the teeth were isolated with rubber dam and access performed. Patients were instructed to definitively rate any pain felt during endodontic procedure. If patient felt pain, the treatment was immediately stopped and the patient rated their discomfort using Heft Parker VAS. The extent of access achieved when the patient felt pain was recorded as within dentin, entering the pulp chamber or initial file placement. The success was defined as the ability to access and instrument the tooth without pain (VAS score of zero) or mild pain (VAS rating<54mm).

DETAILED DESCRIPTION:
The present clinical study was carried out to compare the anaesthetic success of 4% articaine with 2% lidocaine for intraligamentary anaesthesia in patients having irreversible pulpitis.

Subjects randomly received two intraligamentary injections using Ligaject at a two separate appointments spared one week apart in a cross over design. Twenty patients received intraligamentary injections of 0.9 ml of 4%articaine with 1:100,000 epinephrine (Septodont INC) at first appointment and 1.8 ml of lidocaine with 1:100,000 epinephrine. Each patient served as her own control. All injections were given by the same physician or author. The injection was performed by inserting the needle at the gingival sulcus at the mesio-buccal line angle of the tooth with needle directed at approximately 30degrees angle to the long axis of the tooth in the buccolingual plane. Needle was placed into the sulcus with the bevel placing away from the tooth and towards the alveolar bone. Needle was advanced with a firm pressure until it could be advanced no further.

The operator waited 10 seconds before slowly removing the needle from the injection site. This step supposedly allows the anaesthetic solution to dissipate within the tissue and reduces the amount of anaesthetic solution to dissipate within the tissue and reduces the amount of solution dripping from the site before needle withdrawal. However, in almost all cases some anaesthetic solution escaped upon removal of needle from the sulcus.

Five minutes post injection, the teeth were isolated under rubber dam isolation and investigator performed the access cavity. Patients were instructed to definitely rate any pain felt during endodontic procedure. If patient felt pain, the treatment was immediately stopped and the patient rated her discomfort using Heft Parker VAS. The extent of access achieved when the patient felt pain was recorded as within dentin, entering the pulp chamber or initial file placement. The success was defined as the ability to access and instrument the tooth without pain (VAS score of zero) or mild pain (VAS rating<54mm).

ELIGIBILITY:
Inclusion Criteria:

* Irreversible pulpitis in the bilateral first or second mandibular molars.
* Absence of periapical radiolucency on the periapical radiographs(except for periapical widening) confirmed the presence of irreversible pulpitis in the teeth.

Exclusion Criteria:

* Pregnant women,
* Patients with systemic disease .
* Teeth with Previous endodontic therapy, large restorations, full crowns, periodontal diseases, or restoration with poor margins were eliminated from the study.
* Also teeth with a history of trauma or sensitivity were eliminated.
* Patients taken antibiotics or analgesics in previous 3 months

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Pain scale as measured by The Heft Parker Visual scale (HP-VAS) | baseline
  HP-VAS was a 170mm line divided into different categories of pain. Different marks on the line show a description of a certain pain level. Absence of pain corresponded to 0mm. mild pain with the descriptors of faint, weak, and mild pain corresponded to 0mm to 54mm, Moderate pain corresponded to greater than 54mm upto 114mm, and Severe pain with the descriptors of strong, intense, and maximum possible amount of pain corresponded to greater than 114mm upto 170mm. Patients were asked to rate their initial pain on a HP-VAS,

REFERENCES:
- [Background] Malamed SF, Gagnon S, Leblanc D. A comparison between articaine HCl and lidocaine HCl in pediatric dental patients. Pediatr Dent. 2000 Jul-Aug;22(4):307-11. PMID 10969438
- [Background] Vahatalo K, Antila H, Lehtinen R. Articaine and lidocaine for maxillary infiltration anesthesia. Anesth Prog. 1993;40(4):114-6. PMID 7943919